CLINICAL TRIAL: NCT00147264
Title: A Randomized, Double Blind, 2X2 Factorial Design Study to Evaluate the Effects of Telmisartan vs Placebo, and of a Low-Glycemic Diet vs Control Diet, in Reducing Intra-Myocellular Lipids In Individuals With Abdominal Obesity
Brief Title: Telmisartan-Induced Reduction in Intra-Myocellular Lipids Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Boehringer Ingelheim (Industry); Canadian Institutes of Health Research (CIHR) (Other Government); Heart and Stroke Foundation of Canada (Other); Medtronic (Industry)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 502.433; BI Pharmaceuticals - 502.433; CIHR - 116099
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-12

CONDITIONS: Metabolic Syndrome X
Keywords: insulin resistance, myocellular lipids, adipose tissue
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance | interventions — Telmisartan

INTERVENTIONS:
Drug: Telmisartan (Micardis®) vs. Placebo
Behavioral: Low-Glycemic Index Diet vs. Control Diet

SUMMARY:
The purpose of this study is to determine whether telmisartan and/or a low-glycemic index diet are effective in reducing intra-myocellular lipid (muscle fat) content.

DETAILED DESCRIPTION:
The metabolic syndrome currently affects over 20% of the adult population in Canada. Patients with abdominal obesity are at markedly increased risk for diabetes and heart disease. Recent studies have shown that decreased sensitivity to insulin (insulin resistance), a hallmark of the metabolic syndrome, is related to increased storage of fat in muscle cells (muscle fat). Several recent studies indicate that blocking the renin-angiotensin system (RAS) may improve insulin sensitivity and prevent the development of type 2 diabetes. Other data suggests that this effect may be due to the effect of RAS blockade on the recruitment and growth of adipose tissue. The primary aim of this study is therefore to explore the role of angiotensin II in the development of insulin resistance. Specifically, we will examine the mechanisms underlying the putative anti-diabetic effect of RAS blockade by examining the effect of angiotensin receptor blockade on muscle fat content in individuals with the abdominal obesity. This study will therefore test the hypothesis that treatment with the angiotensin receptor blocker telmisartan (Micardis®) will reduce muscle fat, thereby improving insulin sensitivity in people with abdominal obesity, with or without additional features of the metabolic syndrome. A number of dietary factors can also affect insulin sensitivity and may influence muscle fat. Recent studies suggest that increasing the content of low-glycemic foods (carbohydrates which are less easily digested), can improve insulin sensitivity and lipid profile in patients with insulin resistance. A second aim of this study is therefore to test the hypothesis that a low-glycemic diet will reduce muscle fat, thereby improving insulin sensitivity in this population.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Between 30 and 70 years of age
* Abdominal obesity defined as increased waist circumference (Men >102cm (>40in), Women >88cm (>35in)), with or without any of the following additional criteria of the metabolic syndrome:
* Triglycerides >=1.7mmol/L (>=150 mg/dL and/or on prescribed lipid lowering medication for > 3 months)
* HDL cholesterol
* Men <1.0 mmol/L (<40 mg/dL)
* Women <1.3 mmol/L (<50 mg/dL)
* Blood pressure >=130 and/or >=85 mmHg and/or on anti-hypertensive therapy (except ACE-I or ARB)
* Fasting glucose >=6.1 mmol/L (>=110 mg/dL)
* Ability and willingness to complete dietary and activity diaries and questionnaires.

Exclusion Criteria:

* Participant has taken ACE inhibitor or ARB in the last 3 months, or in the opinion of the study physician currently has indication for either of these medications
* Concurrent antidiabetic medication
* Use of systemic glucocorticosteroids (topical and inhaled are acceptable)
* On lipid-lowering medication and NOT on stable dose for the last three months
* If the participant has any one or more of the following medical disorders:

  1. diabetes mellitus and/or FBG >=7.0 mmol/L on two separate occasions within the screening period
  2. uncontrolled hypertension (SBP >=160 mmHg and/or DBP >=100 mmHg) or known participants with secondary causes of hypertension
  3. biliary obstruction
  4. hepatic dysfunction as defined by SGPT (ALT) > 3 times the upper limit of normal range
  5. renal dysfunction as defined by serum creatinine > 130umol/L AND/OR proteinuria 1+ or greater (dipstick)
  6. serum triglycerides >10 mmol/L
  7. history of hypertrophic obstructive cardiomyopathy, hemodynamically relevant stenosis of the aortic or mitral valve
  8. sodium depletion or hyperkalemia.
  9. uncorrected volume depletion
  10. endocrine disorder (e.g. hyperthyroidism, Cushing's syndrome, acromegaly, etc.) Participants on thyroid-replacement therapy and TSH < 5.0 mU/L may be enrolled in the study.
  11. contraindications to study diet
  12. any major surgery that is, at the time of screening, planned to take place during the study period.
  13. previously angioedema with ACE Inhibitor or ARB or known hypersensitivity to any component of the study drug formulations (e.g. hereditary fructose intolerance)
  14. history of drug or alcohol dependency within six months prior to signing the informed consent form.
  15. history of active malignancy, chronic inflammatory disorder, or chronic infections which would interfere with protocol completion.
  16. any other medical, social or geographic condition, which, in the opinion of the investigator would not allow safe completion of the protocol and/or safe administration of trial medication
* If the participant has any contraindications to MRI
* Pre-menopausal women (last menstruation >=1 year prior to consent) who:

  1. are not surgically sterile or
  2. are nursing, or pregnant, or
  3. are of child-bearing potential and are NOT practicing acceptable methods of birth control, or do NOT plan to continue practicing an acceptable method throughout the study, AND do not agree to periodic pregnancy testing during participation in the study.
* Intention to go on weight - reducing medications or weight-loss diets during the study period
* Significant fluctuations in weight over past 3 months(e.g. >10%)
* Household member currently in study
* Any investigational drug therapy within one month of signing the informed consent form.
* Participant has knowledge that he/she will be unable to consume study foods for >2 weeks during treatment phase of study
* <70% compliant during run-in
* Unable to reduce total fat consumption to <40% and/or reduce saturated fat consumption to <15% during run-in

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2004-04; Primary Completion 2006-01 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
(for both interventions): change in IMCL content in the soleus muscle as assessed by 1H-MRI Spectroscopy at baseline and 6 months

SECONDARY OUTCOMES:
Change in intra-hepatocellular lipid storage as assessed by 1H-MRI Spectroscopy
Change in insulin sensitivity as determined by HOMA index
Reversal of IFG to normal fasting glucose in participants with IFG
Change in 72-hour subcutaneous glucose profile
Change in fasting lipid profile (free fatty acids, triglyceride, total cholesterol, low-density lipoprotein (LDL) and high-density lipoprotein (HDL) cholesterol)
Change in serum/plasma levels of inflammatory markers (C-reactive protein, adiponectin, tumor necrosis factor a, interleukin 6, leptin, adhesion molecules, plasminogen-activation inhibitor-1, t-PA, global test of fibrinolysis, fibrinogen, homocysteine,
Change in beta-cell function as assessed by the Insulin Secretion Index
Other efficacy parameters of the AT1 blockade and LGI diet are:
Change in waist circumference
Change in body composition as assessed by bioelectrical impedance analysis
Change in abdominal (visceral) adipose tissue as assessed by MRI
Change in resting blood pressure
Change in adipocytic cell size determined by grouped diameter distribution in subcutaneous abdominal adipose tissue biopsies
Changes in mRNA expression of genes in adipose tissue for genes involved in adipose tissue differentiation, growth, metabolism, cardiovascular function and inflammation.
Change in muscle triglyceride content (histochemical examination of muscle biopsies)
Change in molecular markers of endoplasmic reticular stress in circulating blood cells
Endothelial function as assessed by Doppler ultrasound of the forearm blood flow.
Systolic and diastolic cardiac function as assessed by echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Arya M Sharma, MD, FRCPC, Principal Investigator — McMaster University
Locations (1):
- Hamilton Health Sciences - Cardiovascular Obesity Research and Management Center, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Chetty VT, Damjanovic S, Gerstein H, Singh N, Yusuf S, Anand SS, Sharma AM. Metabolic effects of telmisartan in subjects with abdominal obesity: a prospective randomized controlled trial. Blood Press. 2014 Feb;23(1):54-60. doi: 10.3109/08037051.2013.791411. Epub 2013 Jun 3. PMID 23731019
- [Derived] Kochan AM, Wolever TM, Chetty VT, Anand SS, Gerstein HC, Sharma AM. Glycemic index predicts individual glucose responses after self-selected breakfasts in free-living, abdominally obese adults. J Nutr. 2012 Jan;142(1):27-32. doi: 10.3945/jn.111.146571. Epub 2011 Nov 16. PMID 22090469